CLINICAL TRIAL: NCT00747877
Title: Myeloma X Relapse (Intensive): A Phase III Study to Determine the Role of a Second Autologous Stem Cell Transplant as Consolidation Therapy in Patients With Relapsed Multiple Myeloma Following Prior High-dose Chemotherapy and Autologous Stem Cell Rescue.
Brief Title: High-Dose Melphalan and a Second Stem Cell Transplant or Low-Dose Cyclophosphamide in Treating Patients With Relapsed Multiple Myeloma After Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: LCC-HM05/7287; CDR0000612567 (Registry Identifier: PDQ (Physician Data Query)); EU-20873; ISRCTN60123120; EudraCT-2006-005890-24
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; stage I multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; Melphalan

ARMS (2):
- Arm I (Experimental): Patients receive high-dose melphalan IV on day -1 followed by autologous stem cell transplantation (ASCT) on day 0.
  Interventions: Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation
- Arm II (Experimental): Patients receive low-dose cyclophosphamide IV or orally once a week for 12-20 weeks for a total of 12 courses.
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide — Given orally
  Arms: Arm II
Drug: melphalan — Given IV
  Arms: Arm I
Procedure: autologous hematopoietic stem cell transplantation — Patients undergo autologous hematopoietic stem cell transplantation on day 0.
  Arms: Arm I

SUMMARY:
RATIONALE: Giving chemotherapy and bortezomib before a peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and bortezomib. It is not yet known whether high-dose melphalan given together with a second stem cell transplant is more effective than low-dose cyclophosphamide in treating patients with relapsed multiple myeloma.

PURPOSE: This randomized phase III trial is studying giving high-dose melphalan together with a second stem cell transplant to see how well it works compared with low-dose cyclophosphamide in treating patients with relapsed multiple myeloma after chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect on freedom from disease progression in patients with relapsed multiple myeloma treated with re-induction therapy comprising bortezomib, doxorubicin hydrochloride, and dexamethasone (PAD) followed by a second autologous stem cell transplantation (ASCT) with high-dose melphalan vs low-dose cyclophosphamide consolidation therapy.

Secondary

* To assess the response rate of PAD in patients following a previous autograft.
* To compare the overall response rate of patients following high-dose melphalan chemotherapy and autologous stem cell transplantation with low-dose cyclophosphamide consolidation therapy.
* To assess the overall survival of patients treated with this regimen.
* To assess the safety and toxicity of a second ASCT in these patients.
* To assess the safety and toxicity of PAD in these patients.
* To assess the feasibility of stem cell collection following PAD in these patients.
* To determine the impact of this regimen on pain and quality of life in these patients.

OUTLINE: This is a multicenter study.

* Re-induction (PAD) therapy: Patients receive bortezomib IV on days 1, 4, 8, and 11, doxorubicin hydrochloride IV continuously on days 1-4, and oral dexamethasone on days 1-4 (and days 8-11 and 15-18 of course 1 only). Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Peripheral blood stem cell (PBSC) mobilization and harvest: Within 6-12 weeks, some patients receive cyclophosphamide IV on day 0 and filgrastim (G-CSF) subcutaneously (SC) beginning on day 1 and continuing to time of PBSC harvest. PBSCs are then collected.

Patients who successfully complete re-induction therapy and have adequate PBSC mobilization are stratified according to length of first remission or plateau (≤ vs ≥ 24 months) and response to PAD re-induction therapy (stable disease vs ≥ partial response). Patients are randomized to 1 of 2 arms.

* Arm I (high-dose melphalan consolidation therapy): Patients receive high-dose melphalan IV on day -1 followed by autologous stem cell transplantation (ASCT) on day 0.
* Arm II (low-dose cyclophosphamide consolidation therapy): Patients receive low-dose cyclophosphamide IV or orally once a week for 12-20 weeks for a total of 12 courses.

Patients complete the EORTC QLQ-C30 and EORTC QLQ-MY20, the Brief Pain Inventory Short Form (BPI-SF), and the Leeds Assessment of Neuropathic Symptoms and Signs (Self Assessment) Pain Scale (S-LANSS) questionnaires at baseline and after completion of re-induction therapy.

Patients are followed monthly for up to 100 days after ASCT or at 30 days after low-dose cyclophosphamide and then every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed multiple myeloma

  * Symptomatic disease, including non-secretory
* Previously treated with standard chemotherapy and autologous stem cell transplantation
* Requires therapy for first progressive disease AND at least 18 months since first stem cell transplantation

  * Patients who were previously immunofixation-negative and are now immunofixation-positive must have > 5 g/L absolute increase in paraprotein
* Registered in the Myeloma X Relapse (Intensive) Trial and received 2-4 courses of PAD re-induction chemotherapy according to the protocol (consolidation phase)
* Adequate stem cell mobilization available for transplantation defined as ≥ 2x10^6 CD34 + cells/kg or ≥ 2x10^8 PBMC/kg including cells stored from a previous harvest (consolidation phase)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1 x 10^9/L
* Platelet count ≥ 50 x 10^9/L
* Creatinine clearance ≥ 30 mL/min
* Total bilirubin < 2 times upper limit of normal (ULN)
* ALT or AST < 2.5 times ULN
* History of pulmonary disease allowed provided carbon monoxide diffusion in the lungs (KCO/DLCO) is ≥ 50% and/or no requirement for supplementary continuous oxygen
* Left ventricular ejection fraction ≥ 40% by ECG or MUGA scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No known HIV or Hepatitis B or C positivity (testing is not required)
* No known resistance to combined bortezomib, doxorubicin hydrochloride, and dexamethasone therapy
* No known history of allergy to compounds containing boron or mannitol
* No other previous or concurrent malignancies except for appropriately treated localized epithelial skin cancer or carcinoma in situ of the cervix, or remote histories of other cured tumors within the past 5 years
* No medical or psychiatric condition which, in the opinion of the investigator, contraindicates the patient's participation in the study
* No other contra-indication to treatment that would make the patient ineligible for consolidation phase

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other prior therapy for relapsed disease except for local radiotherapy, therapeutic plasma exchange, or ≤ 200 mg of dexamethasone

  * Radiotherapy since prior transplantation sufficient to alleviate or control pain of local invasion is permitted
* No hemi-body radiation since prior transplantation (consolidation phase)
* At least 4 weeks since prior and no concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2008-04; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression

SECONDARY OUTCOMES:
Response rate to bortezomib, doxorubicin hydrochloride, and dexamethasone (PAD)
Overall response rate following randomized treatments
Overall survival
Progression-free survival
Toxicity and safety of autologous stem cell transplantation
Toxicity and safety of weekly cyclophosphamide
Toxicity and safety of PAD therapy
Feasibility of stem cell collection
Pain
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cook, MD, PhD, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (53):
- United Kingdom (53):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Frenchay Hospital, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - St. Helier Hospital, Carshalton, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Saint Richards Hospital, Chichester, England
  - Colchester General Hospital, Colchester, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's Hospital, London, England
  - King's College Hospital, London, England
  - St. George's Hospital, London, England
  - University College of London Hospitals, London, England
  - Manchester Royal Infirmary, Manchester, England
  - Christie Hospital, Manchester, England
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, England
  - James Cook University Hospital, Middlesbrough, England
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Rotherham General Hospital, Rotherham, England
  - Salisbury District Hospital, Salisbury, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Musgrove Park Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital, Swansea, Wales

REFERENCES:
- [Derived] de Tute RM, Cook G, Cairns DA, Brown JM, Cavenagh J, Ashcroft AJ, Snowden JA, Yong K, Tholouli E, Jenner M, Hockaday A, Drayson MT, Morris TCM, Rawstron AC, Owen RG. Impact of minimal residual disease (MRD) in salvage autologous stem cell transplantation for relapsed myeloma: results from the NCRI Myeloma X (intensive) trial. Bone Marrow Transplant. 2024 Mar;59(3):431-434. doi: 10.1038/s41409-023-02164-4. Epub 2024 Jan 9. No abstract available. PMID 38195983
- [Derived] Cook G, Ashcroft AJ, Cairns DA, Williams CD, Brown JM, Cavenagh JD, Snowden JA, Parrish C, Yong K, Cavet J, Hunter H, Bird JM, Pratt G, Chown S, Heartin E, O'Connor S, Drayson MT, Hockaday A, Morris TC; National Cancer Research Institute Haemato-oncology Clinical Studies Group. The effect of salvage autologous stem-cell transplantation on overall survival in patients with relapsed multiple myeloma (final results from BSBMT/UKMF Myeloma X Relapse [Intensive]): a randomised, open-label, phase 3 trial. Lancet Haematol. 2016 Jul;3(7):e340-51. doi: 10.1016/S2352-3026(16)30049-7. PMID 27374467
- [Derived] Parrish C, Morris CTCM, Williams CD, Cairns DA, Cavenagh J, Snowden JA, Ashcroft J, Cavet J, Hunter H, Bird JM, Chalmers A, Brown JM, Yong K, Schey S, Chown S, Cook G; National Cancer Research Institute Haemato-Oncology Clinical Studies Group. Stem Cell Harvesting after Bortezomib-Based Reinduction for Myeloma Relapsing after Autologous Transplantation: Results from the British Society of Blood and Marrow Transplantation/United Kingdom Myeloma Forum Myeloma X (Intensive) Trial. Biol Blood Marrow Transplant. 2016 Jun;22(6):1009-1016. doi: 10.1016/j.bbmt.2016.01.016. Epub 2016 Jan 28. PMID 26827659
- [Derived] Cook G, Williams C, Brown JM, Cairns DA, Cavenagh J, Snowden JA, Ashcroft AJ, Fletcher M, Parrish C, Yong K, Cavet J, Hunter H, Bird JM, Chalmers A, O'Connor S, Drayson MT, Morris TC; National Cancer Research Institute Haemato-oncology Clinical Studies Group. High-dose chemotherapy plus autologous stem-cell transplantation as consolidation therapy in patients with relapsed multiple myeloma after previous autologous stem-cell transplantation (NCRI Myeloma X Relapse [Intensive trial]): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Jul;15(8):874-85. doi: 10.1016/S1470-2045(14)70245-1. Epub 2014 Jun 16. PMID 24948586
- [Derived] Michaelis LC, Saad A, Zhong X, Le-Rademacher J, Freytes CO, Marks DI, Lazarus HM, Bird JM, Holmberg L, Kamble RT, Kumar S, Lill M, Meehan KR, Saber W, Schriber J, Tay J, Vogl DT, Wirk B, Savani BN, Gale RP, Vesole DH, Schiller GJ, Abidi M, Anderson KC, Nishihori T, Kalaycio ME, Vose JM, Moreb JS, Drobyski W, Munker R, Roy V, Ghobadi A, Holland HK, Nath R, To LB, Maiolino A, Kassim AA, Giralt SA, Landau H, Schouten HC, Maziarz RT, Mikhael J, Kindwall-Keller T, Stiff PJ, Gibson J, Lonial S, Krishnan A, Dispenzieri A, Hari P; Plasma Cell Disorders Working Committee of the Center for International Blood and Marrow Transplant Research. Salvage second hematopoietic cell transplantation in myeloma. Biol Blood Marrow Transplant. 2013 May;19(5):760-6. doi: 10.1016/j.bbmt.2013.01.004. Epub 2013 Jan 5. PMID 23298856